CLINICAL TRIAL: NCT04694391
Title: Genomic Study of Relapse Esophageal Cancer After Radiotherapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Collaborators: M.D. Anderson Cancer Center (Other); Nantong University (Other); Jiangsu Cancer Institute & Hospital (Other); Henan Cancer Hospital (Other Government); Ningbo No.2 Hospital (Other); Taihe Hospital (Other); Taian Cancer Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ESO-shanghai 6
Record Dates: First submitted 2020-12-31; First posted 2021-01-05 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Gene Mutation-Related Cancer; Esophageal Cancer; Radiation Exposure
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA was extracted from all samples to conduct exome sequence. The investigators attempt to seek genomic characteristics of relapsed esophageal cancer after radiotherapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Recurrence: The period of recurrence was within 2 years after radiotherapy. Pathologic diagnosis was squamous cell carcinoma same with preradiotherapy.
  Interventions: Genetic: whole exome sequence
- No recurrence: The period was more than 3 years after radiotherapy and no recurrence signs were observed.
  Interventions: Genetic: whole exome sequence

INTERVENTIONS:
Genetic: whole exome sequence — To seek genomic characteristics of relapsed esophageal cancer with whole exome sequence.

SUMMARY:
Radiotherapy plays an important role in multidisciplinary treatment of esophageal cancer. However, about half patients received radiotherapy occurred relapse. Once relapse occurred, there is no better treatment strategy. Genomic study of relapsed esophageal cancer is seldom. So the investigators attempt to collect relapsed tissue to conduct with whole exome sequencing in order to investigate the genome landscape of recurrence esophageal cancer.

DETAILED DESCRIPTION:
Tumor tissue of patients received radiotherapy with diagnosis of recurrence between Jan 1, 2010 and Dec 1, 2020 were collected retrospectively. Recurrence tumor tissue is collected between Dec 31, 2020 and Dec 31, 2022 prospectively. Blood and preradiotherapy tumor tissue were also collected to be as contrast. A total of 100 paired blood, preradiotherapy tumor tissue and relapse tumor tissue were collected. What is more, a total of 100 paired blood and preradiotherapy tumor tissue with diagnosis of no recurrence were collected. All samples were conducted with whole exome sequencing.

Here the investigators define recurrence period as within 2 years and no recurrence period as more than 3 years after radiotherapy.

Criteria of relapse: (1) pathologic diagnosis is squamous carcinoma before radiotherapy;(2) received radiotherapy; (3)pathologic diagnosis is also squamous carcinoma after radiotherapy; (4) clinical symptoms including feeding obstruction etc; (5) imaging evidence showed disease progression.

ELIGIBILITY:
Inclusion Criteria:

1. pathologic diagnosis is squamous cell carcinoma before radiotherapy;
2. pathologic diagnosis is squamous cell carcinoma after radiotherapy;
3. received radiotherapy
4. clinical symptoms including dysphagia, feeding obstruction, etc
5. image evidence showed disease progression
6. the period of recurrence was within 2 years after radiotherapy

Exclusion Criteria:

1. pathologic diagnosis is not squamous cell carcinoma before radiotherapy;
2. pathologic diagnosis is not squamous cell carcinoma after radiotherapy
3. not received radiotherapy
4. the period of recurrence was more than 2 years after radiotherapy
5. the period of no recurrence was within 3 years after radiotherapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Recurrence group: 100 paired relapsed tumor tissue,blood and preradiotherapy tumor tissue within 2 years after radiotherapy were collected.
  No recurrence group:100 paired blood and preradiotherapy tumor tissue with more than 3 years after radiotherapy were collected
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2012-09-14 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
genomic characteristics of relapsed esophageal cancer | through study completion, an average of 1 year
  gene mutations, copy number variants

CONTACTS AND LOCATIONS:
Overall Officials: Kuaile Zhao, doctor, Principal Investigator — Fudan University
Locations (1):
- Fudan university shanghai cancer center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No